CLINICAL TRIAL: NCT03263910
Title: Phase Ⅲ Placebo-controlled Study of NPO-11 in Chinese Patients Undergoing Gastrointestinal Endoscopy
Brief Title: Study of NPO-11 in Patients Undergoing Gastrointestinal Endoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nihon Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: NPO-11_301
Record Dates: First submitted 2017-08-21; First posted 2017-08-28 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Patients Undergoing Gastrointestinal Endoscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NPO-11 (Experimental)
  Interventions: Drug: NPO-11
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NPO-11 — 20 ml NPO-11
  Arms: NPO-11
Drug: Placebo — 20 ml NPO-11(Placebo)
  Arms: Placebo

SUMMARY:
Chinese patients who require gastrointestinal endoscopy will receive an intra-gastric single dose of NPO-11 20ml. The superiority of NPO-11 compared to placebo as a premedication for endoscopy will be verified in a randomized, double-blind, parallel-assignment design based on the proportion of patients having no gastric peristalsis.

The safety of NPO-11 will be evaluated based on adverse events and adverse drug reactions observed between informed consent and 7 days after administration in comparison with the placebo group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are capable of understanding and complying with protocol requirements in the opinion of the investigator or the sub-investigator.
2. Patients who are able to fill in the informed consent form.
3. Patients who require gastrointestinal endoscopy using a scope of 9mm or greater diameter for follow-up of confirmed or investigation of a suspected upper gastrointestinal disease. (except for transnasal endoscopy and emergency endoscopy)
4. Male or female chinese patients aged _18_ to _80
5. Patients who agree to use routinely adequate contraception from signing of informed consent to follow-up.

Exclusion Criteria:

1. Patients have received any investigational drug of other study within 120 days prior to providing their informed consent.
2. Patients had been administered NPO-11 in the past.
3. Patients who are the study site investigator or sub-investigator, an immediate family member (eg, spouse,parent, child, sibling), or may consent under duress.
4. Patients have a history of upper gastrointestinal tract surgery.
5. Patients have gastric stenosis or deformity that would make observation of peristaltic movement difficult.
6. Patients have bleeding in the upper gastrointestinal tract and require hemostatic intervention.
7. Patients have reflux esophagitis (defined as Los Angeles Class: B, C or D)
8. Patients have an active gastric or duodenal ulcer (defined as Sakita-Miwa class: A1 or A2)
9. Patients are on treatment (radiotherapy or chemotherapy) for cancer.
10. Patient have decreased heart function (NYHA heart function class: III or more)
11. Patients have a history of shock, hypersensitivity or allergies to l-menthol or peppermint oil.
12. Patients have a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 12 months prior to the screening visit.
13. Patients are required to take excluded medications.
14. If female, patients are pregnant or lactating or intending to become pregnant from signing of informed consent to follow-up.
15. Any subject who, in the opinion of the investigator or the sub-investigator, is unable to comply with the requirements of the study or is unsuitable for any reason.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-08-17 (Actual)

PRIMARY OUTCOMES:
The proportion of patients had no gastric peristalsis during the procedures | 15 minutes
  No gastric peristalsis is defined as when patients have no gastric peristalsis at both 2 minutes post-dose and the end of endoscopy.(central evaluation by independent evaluator)

SECONDARY OUTCOMES:
Change in peristaltic movement | 15 minutes
  The measure use peristaltic grade(central evaluation by independent evaluator).
Difficulty level of intra-gastric observation | 15 minutes
  Subjective evaluation by investigator or subinvestigator who performs endoscopy
Correlation between the time from the dose to the end of endoscopy and peristaltic grade | 15 minutes

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - East China, East China
  - North China
  - Northwest China
  - South China

REFERENCES:
- [Derived] Meng F, Li W, Zhi F, Li Z, Xue Z, He S, Chen W, Chen Y, Xing X, Yao C, Wu Y, Zhang S. Antiperistaltic effect and safety of l-menthol oral solution on gastric mucosa for upper gastrointestinal endoscopy in Chinese patients: Phase III, multicenter, randomized, double-blind, placebo-controlled study. Dig Endosc. 2021 Nov;33(7):1110-1119. doi: 10.1111/den.13941. Epub 2021 Apr 2. PMID 33527576